CLINICAL TRIAL: NCT05596370
Title: Confirmation of Association Between Cell-free Nucleic Acid in Blood and Urine Samples and Microbiome in Stool With Pancreatobiliary Cancer and Study Related to Exploration of Biomarkers in Diagnosis and Treatment of Pancreatobiliary Cancers
Brief Title: Association Between Cell-free Nucleic Acid in Blood, Urine and Microbiome in Stool With Pancreatobiliary Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: DXOME CO., LTD. (Unknown)
Responsible Party: Principal Investigator, Sang Hyub Lee, Professor, Seoul National University Hospital
Other Study IDs: H-2111-199-1281
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Pancreatic Cancer; Cholangiocarcinoma; Gallbladder Cancer
Keywords: cell-free nucleic acid; microbiome; biomarker
MeSH Terms: conditions — Pancreatic Neoplasms; Cholangiocarcinoma; Gallbladder Neoplasms | interventions — Blood Specimen Collection; Urination; Microbiota; Defecation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- biliary cancer: cholangiocarcinoma gallbladder cancer
  Interventions: Diagnostic Test: cell free DNA in blood and urine, metabolite/microbiome in urine and stool
- pancreatic tumor: pancreatic cancer pancreatic ductal adenocarcinoma pancreatic neuroendocrine tumor
  Interventions: Diagnostic Test: cell free DNA in blood and urine, metabolite/microbiome in urine and stool

INTERVENTIONS:
Diagnostic Test: cell free DNA in blood and urine, metabolite/microbiome in urine and stool — cell free DNA in blood and urine, metabolite/microbiome in urine and stool

SUMMARY:
Based on the cell free nucleic acid analysis information of blood samples, the results of microbiome and metabolite analysis of stool and urine samples of pancreatic cancer and bile duct cancer patients, the clinical correlations of them with primary cancer are evaluated. And based on these information, biomarkers for diagnosis, treatment, and prognosis of pancreatic and bile duct cancer are explored.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with pancreatic cancer through histological or radiologic examination and before treatment begins
* Patients diagnosed with biliary tract cancer (cholangiocarcinoma, gallbladder cancer) through histological or radiologic examination and before treatment begins
* Patients aged 18 or older who voluntarily agrees to participate in the study and is willing to understand and comply with the subsequent treatment procedures and sample collection schedule

Exclusion Criteria:

* Where the subject himself/herself refuses to fill out the consent form or is unable to fill out the consent form
* In the case where the sample storage conditions suggested by the reagent manufacturer are not satisfied
* Only samples that can cause errors when determining results are acquired:

  * Heat treated specimen

    * Incompletely coagulated serum and bacterial samples ③ Samples with particulate matter elements (e.g., fibroblasts, red blood cells) remaining in the sample

      ④ Specimens previously frozen and stored with blood clots that have confirmed an increase in non-specific reactivity in which samples appear to have denatured during storage

      ⑤ Sample from deceased patient

      ⑥ A patient specimen with a malignancy of ohter site

      ⑦ Sample from vulnerable persons such as pregnant women, minors, etc

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 or older, who diagnosed with pancreatic cancer or biliary tract cancer (cholangiocarcinoma, gallbladder cancer) through histological or radiologic examination and before treatment begins
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-01-06 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
correlation of genetic mutation | the day of study enrollment or the day of tissue and blood acquisition
  concordance of genetic mutation between tissue and blood of treatment-naive status
correlation of genetic mutation burden and prognosis | the day of study enrollment and follow-up till end of the study
  correlation of genetic mutation burden and prognosis

SECONDARY OUTCOMES:
correlation of metabolic change in urine metabolite and prognosis | the day of study enrollment and follow-up till end of the study
  analysis of correlation of metabolic change in urine metabolite and prognosis
correlation of microbiome in stool and prognosis | the day of study enrollment and follow-up till end of the study
  analysis of correlation of microbiome in stool and prognosis

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Sang Hyub Lee, Seoul

IPD SHARING:
Plan to Share IPD: No